CLINICAL TRIAL: NCT07262684
Title: The Effect of the Psychological Resilience Workshop Implemented After the Kahramanmaraş Earthquakes on University Students' Levels of Psychological Resilience
Brief Title: Resilience Training for University Students After the Earthquakes
Acronym: RSUS-AE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Ege Miray Topcu, Researcher, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 424K083; 424K083 (Other: TÜBİTAK)
Record Dates: First submitted 2025-11-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Psychological Resilience; Psychological Well-being
Keywords: psychological resilience; psychogical well-being; Earthquake; university students
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The study is a controlled, single-blind, randomized, experimental follow-up study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention Group (Experimental): A six-session program was implemented with this group. The program was delivered face-to-face in a group format.
  Interventions: Behavioral: Psychological Resilience Workshops
- control group (No Intervention): control: At the time the intervention group completed the program, this group was administered the post-test and follow-up test. No intervention was provided; however, participants were informed at the beginning and end of the study about available psychological support services if needed.

INTERVENTIONS:
Behavioral: Psychological Resilience Workshops — Psychological Resilience Workshops are designed as a comprehensive group program aimed at strengthening university students' levels of psychological resilience and well-being. Grounded in the principles of Cognitive Behavioral Theory, the program is enriched with expressive arts techniques that support emotional awareness and self-expression. Over the course of six weeks, participants engage in activities that foster self-awareness, self-esteem, social support, and flexibility skills, helping them explore and enhance their own psychological resilience. Drawing on research findings emphasizing the importance of self-esteem, well-being, and sense of belonging among university students, the Psychological Resilience Workshops are structured to directly promote these areas.
  Arms: İntervention Group

SUMMARY:
Earthquakes can have strong emotional effects on people, especially large disasters such as the Kahramanmaraş earthquakes on February 6, 2023. The anniversaries of such events can be difficult times when fear, anxiety, and memories of loss may return. This study aims to increase the psychological resilience and psychological well-being of university students who are beginning their first year.

The target group of this study is students in the foreign language preparatory program, whether they have personally experienced the earthquake or not. The study will examine the effects of a six-week workshop program designed for these students.

The study includes three measurement points: a pre-test, a post-test, and a follow-up test. All students will be invited to complete the initial screening, which will assess their resilience and psychological well-being levels. Students who meet the eligibility criteria will be randomly assigned to either the intervention group (18 students) or the control group (18 students).

Students in the intervention group will participate in the Psychological Resilience Workshop, which takes place once a week for six weeks and lasts about 60-90 minutes per session. The workshop combines a cognitive-behavioral approach with creative emotional expression activities. During the sessions, students will work on understanding themselves, recognizing difficult emotions, identifying their sources of support, and strengthening their psychological resilience. Activities include drawing, storytelling, creative exercises, and group games.

Students in the control group will not receive an intervention but will be provided with information about psychological support services they can access if needed.

The workshop is expected to increase students' psychological resilience and psychological well-being in both the short term and the long term. The results of this study may help develop a practical, sustainable, low-cost mental health support program that can be used with university students.

DETAILED DESCRIPTION:
The earthquakes that occurred on February 6, 2023, in Kahramanmaraş were large-scale disasters that directly or indirectly affected individuals across a wide region. The anniversaries of major traumatic events are known to be periods in which anxiety, mood fluctuations, reactivation of loss-related memories, and emotional sensitivity may intensify. This process can be particularly impactful for university students, who are in a developmental stage that involves significant academic, social, and emotional transitions. Regardless of whether they directly experienced the earthquake, first-year language preparatory students represent a heterogeneous group and may display varying levels of psychological impact.

Psychological resilience refers to the capacity to cope with stress, adversity, or trauma while maintaining functional well-being. Strengthening resilience is known to support emotional regulation, adaptability, and effective coping skills. Previous studies indicate that group-based resilience interventions rooted in cognitive-behavioral principles can be beneficial for young adults.

This study is designed as a randomized controlled experimental trial conducted with students enrolled in the university's foreign language preparatory program. In the initial phase, all preparatory students will be invited to participate in an online screening assessment. Students meeting the inclusion criteria will be randomly assigned to the intervention or control group. Randomization will be stratified according to the province in which students resided during the earthquake period, ensuring balanced representation of those who experienced the earthquake and those who did not, thereby improving comparability between groups.

The intervention group will participate in a six-session "Psychological Resilience Workshop," developed based on cognitive-behavioral principles and enhanced with expressive arts techniques. The sessions focus on themes such as self-perception, goal setting, emotional awareness, interpersonal support resources, coping with loss and adversity, and the development of an individualized resilience framework. The program content has been structured with expert consultation. The control group will not receive any intervention but will be provided with information about available support resources should they experience psychological distress.

The study includes three assessment time points: pre-test, post-test, and follow-up. This structure allows for evaluation of both the short-term and medium-term effects of the intervention. The findings are expected to contribute to the development of an accessible, cost-effective, and evidence-based psychological resilience program suitable for university populations.

ELIGIBILITY:
Inclusion Criteria:Voluntary participation

Being over 18 years of age and not having a legal guardian

Attending at least 80% of the workshop sessions

Having sufficient reading ability and physical capacity to complete the data collection form independently -

Exclusion Criteria:Presence of cognitive impairments that prevent completion of the data collection forms (e.g., difficulties in comprehension, speech, reasoning, or decision-making)

Receiving professional psychological support that could affect resilience or well-being during the data collection period

Being officially enrolled in the academic term but not actively attending in-person education

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Connor-Davidson Resilience Scale - Short Form | pretest(around the period after the anniversary of the earthquake), posttest (after workshop), follow test (after four week)
  The Connor-Davidson Resilience Scale was developed by Connor and Davidson (2003) to assess individuals' psychological resilience following adverse life events. The original scale consists of 25 items rated on a 5-point Likert scale ranging from 0 (not true at all) to 4 (true nearly all the time). Psychometric evaluations demonstrated high internal consistency, with a Cronbach's alpha of 0.89 (Connor & Davidson, 2003). Short-form versions were later developed based on factor analytic studies. The Turkish adaptation and psychometric assessment of the short form were conducted by Kaya and Odacı (2021). Higher scores indicate higher levels of psychological resilience. The scale is self-administered and takes approximately five minutes to complete. In the present study, the scale was administered at three time points: pre-test, post-test, and follow-up.
Psychological Well-Being Scale | pretest(around the period after the anniversary of the earthquake), posttest (after workshop), follow test (after four week)
  The Psychological Well-Being Scale was developed by Diener and colleagues (Diener et al., 1985, 2010) and adapted into Turkish by Telef (2013). The scale is used to evaluate individuals' socio-psychological well-being. It consists of 8 items rated on a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree), yielding a total score between 8 and 56. All items are positively worded. As the scale does not include sub-dimensions, higher scores indicate that individuals possess greater psychological resources, such as positive relationships, a sense of competence, and a meaningful and purposeful life. Psychometric studies have demonstrated that the scale is valid and reliable for use with university students in Türkiye (SRMR = 0.04, RMSEA = 0.08, GFI = 0.96, RFI = 0.92, NFI = 0.94, CFI = 0.95, IFI = 0.95). The scale is self-administered and requires approximately five minutes to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Emel Öztürk Turgut, PhD, Study Chair — Ege University
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Analytic Code